CLINICAL TRIAL: NCT01121692
Title: Venue-Based Recruitment and HIV Prevention for Alcohol and Other Drug (AOD) Using Couples in South Africa
Brief Title: Venue-Based Couples CoOp in South Africa
Acronym: Couples CoOp
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: RTI International (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH); Medical Research Council, South Africa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: NIAAA-Wechsberg-AA018076; R01AA018076 (NIH)
Record Dates: First submitted 2010-05-06; First posted 2010-05-12 (Estimated); Last update posted 2015-10-12 (Estimated); Status verified 2015-10

CONDITIONS: Alcoholism; HIV Infections
Keywords: Couples; Alcohol use; HIV risk; Outreach
MeSH Terms: conditions — Alcoholism; HIV Infections; Alcohol Drinking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- VCT/Women's CoOp (Experimental)
  Interventions: Behavioral: Women's CoOp
- Women's CoOp/Men's CoOp (Experimental)
  Interventions: Behavioral: Women's CoOp and Men's Intervention
- Couples CoOp (Experimental)
  Interventions: Behavioral: Couples Intervention

INTERVENTIONS:
Behavioral: Couples Intervention — The Couples intervention is a merged intervention of three interventions (Women CoOp, men as partners's and couples). Couples attend together for two half day workshops and work on exercises on communication and problem solving, including a commitment pledge of fidelity.
  Arms: Couples CoOp
Behavioral: Women's CoOp — The Women's CoOp is a gender-focused intervention discussing women's risk in relationship to HIV and also discusses issues of HIV with South African women including skills for violence prevention. During this intervention, participants will also demonstrate the proper use of male and female condoms on penile and vaginal models. They attend two half day workshops.
  Arms: VCT/Women's CoOp
Behavioral: Women's CoOp and Men's Intervention — The Men's CoOp is adapted from Men as Partners, the Women's CoOp and the Couples intervention and contain similar material with a concentration on gender roles and violence prevention. Men attend two half day workshops.
  Arms: Women's CoOp/Men's CoOp

SUMMARY:
Couples who use alcohol and other drugs (AOD) in South Africa are at high risk for engaging in risky sex behavior within their relationships and with other sexual partners. In addition, high levels of gender-based violence (GBV) in the Cape Town area intersect with AOD abuse and sex behavior. All of these interconnections raise concern for the importance of HIV prevention strategies within or surrounding drinking venues, where many of these behaviors occur.

The specific aims of this study are as follows:

Aim 1. To characterize the types of drinking venues (e.g., licensure status, size, plumbing, type of alcohol provided), their immediate context (e.g., observed availability and use of other drugs, observable violence and sexual activity), and surrounding neighborhood characteristics (e.g., quality of streets, building structures, and availability of electricity and plumbing) in the sampled neighborhood blocks in several large Black/African and Coloured communities in Cape Town, South Africa.

Aim 2. To refine through qualitative methods the proposed interventions in relation to skills-building to address gender-role expectations, sexual partnering, gender and power, violence, and environments where drinking and sexual risk behaviors occur.

Aim 3. To conduct a randomized group trial to compare the relative efficacy of a comprehensive intervention (Condition 3: Enhanced Couples) to the gender-focused intervention (Condition 2: Gender) and to (Condition 1: Men's Control and Women's CoOp) on reducing alcohol and other drug (AOD) use, sexual risk behavior, and gender-based violence at 6 month follow-ups. Aim 4. To assess the mechanisms through which the intervention effects may occur (e.g., mediators involving self-efficacy and condom mastery, negotiation, and communication skills) and to identify groups for whom the interventions have the greatest effect (e.g., partner characteristics such as race, gender, and age and neighborhood factors such as poverty) on study outcomes of AOD use, sexual risk, and gender-based violence.

ELIGIBILITY:
Men

Inclusion:

* Male
* 18-35
* Identify as Black or Coloured
* Live in one of the target communities- Khayelitsha, Mitchell's Plain and Delft
* Have the same main heterosexual sex partner for at least one year, plan to stay with this partner for at least one year and do not plan to get this partner pregnant within the next year
* Report unprotected sex at least once in the past 90 days with main partner
* Have used alcohol in a tavern or shebeen in the past 90 days
* Spend time in a tavern or shebeen at least weekly

Exclusion

* Have been a part of previous Couples' Health CoOp group study activities
* Are currently enrolled in an HIV research study

Women

Inclusion:

* Female
* 18 or older
* Have the same main heterosexual sex partner for at least one year and plan to stay together with this partner for at least one year and do not plan to get pregnant within the next year with this partner
* Report unprotected sex at least once in the past 90 days with main partner

Exclusion:

* Have been a part of previous Couples' Health CoOp group study activities
* Are currently enrolled in an HIV research study
* Have been a part of the Cape Town Pilot Study or the Western Cape Women's Health CoOp

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2010-05; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Reduced alcohol use | 6 month follow up

SECONDARY OUTCOMES:
reduced gender-based violence | 6 month follow up

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Research Council, Cape Town, South Africa

REFERENCES:
- [Background] Browne FA, Wechsberg WM. The intersecting risks of substance use and HIV risk among substance-using South African men and women. Curr Opin Psychiatry. 2010 May;23(3):205-9. doi: 10.1097/YCO.0b013e32833864eb. PMID 20308902
- [Background] Wechsberg WM, Myers B, Reed E, Carney T, Emanuel AN, Browne FA. Substance use, gender inequity, violence and sexual risk among couples in Cape Town. Cult Health Sex. 2013;15(10):1221-36. doi: 10.1080/13691058.2013.815366. Epub 2013 Aug 8. PMID 23927691
- [Background] Minnis AM, Doherty IA, Kline TL, Zule WA, Myers B, Carney T, Wechsberg WM. Relationship power, communication, and violence among couples: results of a cluster-randomized HIV prevention study in a South African township. Int J Womens Health. 2015 May 11;7:517-25. doi: 10.2147/IJWH.S77398. eCollection 2015. PMID 25999767
- [Background] Doherty IA, Myers B, Zule WA, Minnis AM, Kline TL, Parry CD, El-Bassel N, Wechsberg WM. Seek, Test and Disclose: knowledge of HIV testing and serostatus among high-risk couples in a South African township. Sex Transm Infect. 2016 Feb;92(1):5-11. doi: 10.1136/sextrans-2014-051882. Epub 2015 Jul 14. PMID 26175479
- [Background] Wechsberg WM, Doherty IA, Myers B, Morgan-Lopez AA, Emanuel A, Carney T, Kline TL, Zule WA. Contextualizing gender differences and methamphetamine use with HIV prevalence within a South African community. Int J Drug Policy. 2014 May;25(3):583-90. doi: 10.1016/j.drugpo.2013.10.016. Epub 2013 Nov 9. PMID 24316002
- [Background] El-Bassel, N., & Wechsberg, W.M. Couple-based behavioral HIV intervention: Placing HIV risk-reduction responsibility on the female and male dyad. Couple and Family Psychology 1(2) 94-105, 2012. doi:10.1037/a0028890
- [Derived] Speizer IS, Zule WA, Carney T, Browne FA, Ndirangu J, Wechsberg WM. Changing sex risk behaviors, gender norms, and relationship dynamics among couples in Cape Town, South Africa: Efficacy of an intervention on the dyad. Soc Sci Med. 2018 Jul;209:95-103. doi: 10.1016/j.socscimed.2018.05.024. Epub 2018 May 18. PMID 29843074
- [Derived] Wechsberg WM, Zule WA, El-Bassel N, Doherty IA, Minnis AM, Novak SD, Myers B, Carney T. The male factor: Outcomes from a cluster randomized field experiment with a couples-based HIV prevention intervention in a South African township. Drug Alcohol Depend. 2016 Apr 1;161:307-15. doi: 10.1016/j.drugalcdep.2016.02.017. Epub 2016 Feb 18. PMID 26946991
- [Derived] Wechsberg WM, El-Bassel N, Carney T, Browne FA, Myers B, Zule WA. Adapting an evidence-based HIV behavioral intervention for South African couples. Subst Abuse Treat Prev Policy. 2015 Feb 24;10:6. doi: 10.1186/s13011-015-0005-6. PMID 25888856